CLINICAL TRIAL: NCT01404988
Title: VIP (Veterans Intensive Personalized) Treatment in Heart Failure
Brief Title: Veterans Intensive Personalized Treatment in Heart Failure
Acronym: VIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RRP 11-238
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Results first posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Telemedicine; Medication Adherence
MeSH Terms: conditions — Heart Failure; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telephone-Delivered BI (Experimental): Comprehensive behavioral intervention (BI) - Participants will receive the BI that is based on the transtheoretical model, which targets stage of change, decisional balance and self-efficacy, while also assessing and counseling regarding the barriers and facilitators of HF care, and to improve self-regulatory care such as self-monitoring, self-evaluation, feedback and reinforcement.
  Interventions: Behavioral: Telephone-Delivered BI
- Telephone-Delivered BEI (Experimental): Behavioral & Environmental Intervention (BEI) - Participants in this arm will receive the BI but will also receive environmental tailoring. Environmental Tailoring consists of Built Environment Tailoring (BET) where the intervention will incorporate aspects from the patients' environment, such as accessibility of health food stores or recreational facilities. Environmental Tailoring also consists of Human Environment Tailoring (HET) which incorporates patients' social support. Caregivers will be enrolled for patients in this arm of the study and they will also receive health education.
  Interventions: Behavioral: Telephone-Delivered BEI
- Telephone-Delivered API (Placebo Comparator): Attention Placebo Intervention (API) - patients will receive non-tailored counseling on general health topics.
  Interventions: Other: Telephone-Delivered API

INTERVENTIONS:
Behavioral: Telephone-Delivered BI — Behavioral Intervention will be delivered over the phone.
  Arms: Telephone-Delivered BI
Behavioral: Telephone-Delivered BEI — Behavioral and Environmental Intervention will be delivered over the phone
  Arms: Telephone-Delivered BEI
Other: Telephone-Delivered API — Attention Placebo Intervention will be delivered over the phone
  Arms: Telephone-Delivered API

SUMMARY:
In the VIP (Veterans Intensive Personalized) Treatment in Heart Failure Study we will assess 2 novel interventions to enhance adherence and improve quality of life in veterans with heart failure. This 3-arm randomized controlled trial will base one active arm on how ready patients are for change in terms of diet and medication adherence and will tailor the intervention based on this. The other active arm will also assess how ready patients are for change, but will also include tailoring based on availability of environment resources, such as proximity to health food stores or social support, to further tailor the intervention. The last active arm is simply an attention group where patients will receive general health counseling in addition to background care that all patients receive. The overarching hypothesis is that the tailored interventions will lower heart failure (HF) recurrence and improve quality of life by better medication and diet adherence compared to attention placebo.

DETAILED DESCRIPTION:
OBJECTIVES: In the VIP (Veterans Intensive Personalized) Treatment in Heart Failure Study we will assess 2 novel interventions to enhance adherence and improve quality of life (QOL) in veterans with heart failure (HF). This theory-based pilot 3-arm randomized controlled trial (RCT) will base one active arm on the Transtheoretical Model (TTM), while the other active arm will add environmental (built and human) tailoring to TTM. The overarching hypothesis driving this proposal is that a behavioral intervention (BI), which uses the TTM, or a behavioral and environment-tailored intervention (BEI) will lower HF recurrence and improve QOL by better medication and diet adherence compared to attention control.

RESEARCH DESIGN: This is a practice-based RCT to test the effect of BI and BEI on medication and diet adherence. The study is embedded in typical VA healthcare with all 3 arms incorporating the enhancements in HF care that have been implemented including the Patient Aligned Care Teams (PACT), system redesign methods to improve HF care, ongoing HF quality improvement and Telehealth. We will randomize 99 participants equally to BI, BEI and AP. All analyses will be intent to treat.

METHODOLOGY: The study sites will be the VAMC's at Manhattan and Brooklyn. Participants will be veterans with classes I-III HF with prescribed HF medication for 6 months. Men and women ( 21 years) with history and clinical findings of chronic, stable HF of NYHA functional class I (previously symptomatic/now asymptomatic), II, or III are eligible. They must have an available phone and 2 clinic visits in the previous 1.5 years. Patients with poor short-term survival (< 1 year), recent major surgery (< 3 months), temporarily in the area, or those unable to provide consent will be excluded. After being screened for eligibility, participants will come in for 2 study visits over the course of 6 months which will last about 1.5-2 hours. At each visit, a research assistant (RA) will administer a questionnaire assessing health behaviors including diet, exercise and medication and quality of life. The RAs will also measure height, weight, take 6 BP readings, and send patients to the lab for blood and urine samples. After the first clinic visit, participants will be randomized to one of three telephone groups. All participants will receive 1 phone call per month for 6 months which will last approximately 30-40 minutes. 1) The BI group will receive TTM stage-matched counseling. The interventionist will assess how ready patients are for change in terms of diet, medication, and exercise adherence and deliver a tailored intervention discussing adherence barriers. 2) In the BEI, in addition to using the TTM, the intervention will tailor environmental factors, such as availability of healthy food stores, recreational facilities, and support from caregivers in helping participants follow treatment recommendations. We will speak with participant's caregivers to educate them on heart failure as well. The caregivers will receive a call every 2 months (3 in total) lasting approximately 20-30 minutes. 3) The control group will receive monthly telephone calls during which they will receive general health education. Our primary analytic goal is to estimate the medication adherence rate and QOL to power a larger study. We will also perform 1-sample Exact Binomial Tests comparing the active arms to the expected inactive control rate of 47%. Since this is a pilot study, we will use a 5% type 1 error rate (2-sided) for each test. All analyses will be intent to treat.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (21 years) with history and clinical findings of chronic, stable HF of NYHA functional class I (previously symptomatic/now asymptomatic), II, or III.
* They must have an available phone and 2 clinic visits in the previous 1.5 years.

Exclusion Criteria:

* Patients with poor short-term survival (< 1 year)
* recent major surgery (< 3 months)
* temporarily in the area
* or those unable to provide consent will be excluded.
* Patients excluded and reason for exclusion will be recorded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sundar Natarajan, MD MSc, Principal Investigator — VA New York Harbor Health Care System
Locations (1):
- VA New York Harbor Health Care System, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Comprehensive Behavioral Intervention (BI): Participants will receive the BI that is based on the transtheoretical model, which targets stage of change, decisional balance and self-efficacy, while also assessing and counseling regarding the barriers and facilitators of HF care, and to improve self-regulatory care such as self-monitoring, self-evaluation, feedback and reinforcement over the phone.
- Behavioral & Environmental Intervention (BEI): Participants in this arm will receive the BI but will also receive environmental tailoring. Environmental Tailoring consists of Built Environment Tailoring (BET) where the intervention will incorporate aspects from the patients' environment, such as accessibility of health food stores or recreational facilities. Environmental Tailoring also consists of Human Environment Tailoring (HET) which incorporates patients' social support. Caregivers will be enrolled for patients in this arm of the study and they will also receive health education. Behavioral and Environmental Intervention will be delivered over the phone
- Attention Placebo Group (API) -: Patients will receive non-tailored counseling on general health topics. Attention Placebo Intervention will be delivered over the phone
Period: Overall Study
Arm/Group | Comprehensive Behavioral Intervention (BI) | Behavioral & Environmental Intervention (BEI) | Attention Placebo Group (API) -
Started | 33 | 33 | 33
Completed | 27 | 29 | 30
Not Completed | 6 | 4 | 3
Not completed — Death | 2 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Comprehensive Behavioral Intervention (BI): Participants will receive the BI that is based on the transtheoretical model, which targets stage of change, decisional balance and self-efficacy, while also assessing and counseling regarding the barriers and facilitators of HF care, and to improve self-regulatory care such as self-monitoring, self-evaluation, feedback and reinforcement.Behavioral Intervention will be delivered over the phone.
- Behavioral and Environmental Intervention (BEI): Participants in this arm will receive the BI but will also receive environmental tailoring. Environmental Tailoring consists of Built Environment Tailoring (BET) where the intervention will incorporate aspects from the patients' environment, such as accessibility of health food stores or recreational facilities. Environmental Tailoring also consists of Human Environment Tailoring (HET) which incorporates patients' social support. Caregivers will be enrolled for patients in this arm of the study and they will also receive health education. Behavioral and Environmental Intervention will be delivered over the phone
- Attention Placebo Intervention (API): Patients will receive non-tailored counseling on general health topics. Attention Placebo Intervention will be delivered over the phone
- Total: Total of all reporting groups
Arm/Group | Comprehensive Behavioral Intervention (BI) | Behavioral and Environmental Intervention (BEI) | Attention Placebo Intervention (API) | Total
Number analyzed (Participants) | 33 | 33 | 33 | 99
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65.9 [54.7 to 69.9] | 67.7 [64.5 to 79.1] | 67.6 [64.1 to 75.8] | 67.0 [62.3 to 77.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 32 | 33 | 33 | 98
Race/Ethnicity, Customized [Number; unit: participants]
  White (Non-Hispanic) | 14 | 14 | 16 | 44
  Black (Non-Hispanic) | 13 | 9 | 14 | 36
  Hispanic | 4 | 8 | 1 | 13
  Other | 2 | 2 | 2 | 6
Marital Status [Number; unit: participants]
  Married | 25 | 16 | 25 | 66
  Not Married | 8 | 17 | 8 | 33
Education [Number; unit: participants]
  High School Graduate or Below | 3 | 4 | 2 | 9
  Some College or Higher | 30 | 29 | 31 | 90
Employment Status [Number; unit: participants]
  Employed | 2 | 5 | 5 | 12
  Not Employed | 31 | 28 | 28 | 87
Campus [Number; unit: participants]
  Manhattan | 14 | 12 | 13 | 39
  Brooklyn | 19 | 21 | 20 | 60
Ischemic Heart Disease (IHD) [Number; unit: participants] — Self-reported history
  participants
    History of IHD | 0 | 1 | 1 | 2
    No History of IHD | 33 | 32 | 32 | 97
Medication Adherence [Number; unit: participants] — Self-reported adherence assessed using the Morisky Scale. A score of 0 was classified as high adherence, scores ranging from 1-2 were classified as medium adherence, and scores ranging from 3-8 were classified as low adherence.
  participants
    Low adherence | 5 | 9 | 4 | 18
    Medium Adherence | 15 | 15 | 15 | 45
    High Adherence | 13 | 9 | 14 | 36
Number of Heart Failure Medications [Median (Inter-Quartile Range); unit: number of heart failure medications] | 3.0 [2.0 to 4.0] | 3.0 [3.0 to 4.0] | 3.0 [3.0 to 4.0] | 3.0 [3.0 to 4.0]
Prescribed ACE inhibitors or Angiotensin II Receptor Blockers (ABRs) [Number; unit: participants]
  Prescribed ACE and/or ARB | 23 | 25 | 31 | 79
  Not prescribed ACE and/or ARB | 10 | 8 | 2 | 20
Prescribed Beta Blockers [Number; unit: participants]
  Prescribed Beta Blockers | 32 | 31 | 28 | 91
  Not prescribed Beta Blockers | 1 | 2 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence (Refill Compliance for All HF Medications)
Description: Refill compliance is an objective measurement of medication adherence that utilizes pharmacy records to assess the proportion of time a patient has medication available to take. At the original release of the medication, and each subsequent refill, individuals are given enough medication to last a set number of days. This number is referred to as the "Days Supply" and can be calculated by dividing the number of pills prescribed by the number of pills taken per day. To calculate compliance, the "Days Supply" is subtracted by the number of days between Actual Refill dates, a time span referred to as the "Days Passed". If the Days Passed exceeds the Days Supply the absolute value of the difference represents the number of days the individual was non-adherent. This absolute value is referred to as a "Gap". The sum of the Gaps/total number of days passed between the original release of the medication and the final recorded refill date represents non-compliance over that period of time.
Time Frame: 6 months from baseline visit
Measure: Median (Inter-Quartile Range); unit: proportion of refill compliance
Groups:
- Comprehensive Behavioral Intervention (BI) -: Participants will receive the BI that is based on the transtheoretical model, which targets stage of change, decisional balance and self-efficacy, while also assessing and counseling regarding the barriers and facilitators of HF care, and to improve self-regulatory care such as self-monitoring, self-evaluation, feedback and reinforcement.
  Behavioral Intervention will be delivered over the phone.
- Behavioral & Environmental Intervention (BEI): Participants in this arm will receive the BI but will also receive environmental tailoring. Environmental Tailoring consists of Built Environment Tailoring (BET) where the intervention will incorporate aspects from the patients' environment, such as accessibility of health food stores or recreational facilities. Environmental Tailoring also consists of Human Environment Tailoring (HET) which incorporates patients' social support. Caregivers will be enrolled for patients in this arm of the study and they will also receive health education.Behavioral and Environmental Intervention will be delivered over the phone
- Attention Placebo Group (API): Patients will receive non-tailored counseling on general health topics. Attention Placebo Intervention will be delivered over the phone
Arm/Group | Comprehensive Behavioral Intervention (BI) - | Behavioral & Environmental Intervention (BEI) | Attention Placebo Group (API)
Number analyzed (Participants) | 30 | 29 | 29
proportion of refill compliance | 0.94 [0.86 to 0.99] | 0.97 [0.82 to 1.0] | 0.99 [0.89 to 1.0]
Statistical Analysis 1: Comparison: Comprehensive Behavioral Intervention (BI) - vs Attention Placebo Group (API); Test type: Superiority or Other; p = 0.1, Wilcoxon (Mann-Whitney) — For this pilot study, the Type 1 error was set at 5%
Statistical Analysis 2: Comparison: Behavioral & Environmental Intervention (BEI) vs Attention Placebo Group (API); Test type: Superiority or Other; p = 0.2, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Adherence to ACE Inhibitors and ARB
Description: as for outcome 1
Time Frame: 6 months after baseline
Measure: Median (Inter-Quartile Range); unit: proportion of refill compliance
Groups:
- Comprehensive Behavioral Intervention (BI): Participants will receive the BI that is based on the transtheoretical model, which targets stage of change, decisional balance and self-efficacy, while also assessing and counseling regarding the barriers and facilitators of HF care, and to improve self-regulatory care such as self-monitoring, self-evaluation, feedback and reinforcement. Behavioral Intervention will be delivered over the phone.
Arm/Group | Comprehensive Behavioral Intervention (BI) | Behavioral & Environmental Intervention (BEI) | Attention Placebo Group (API)
Number analyzed (Participants) | 24 | 20 | 25
proportion of refill compliance | 0.98 [0.82 to 1.0] | 1.0 [0.88 to 1.0] | 1.0 [0.99 to 1.0]
Statistical Analysis 1: Comparison: Comprehensive Behavioral Intervention (BI) vs Attention Placebo Group (API); Test type: Superiority or Other; p = .3, Wilcoxon (Mann-Whitney) — For this pilot study, the type 1 error was set at 5%
Statistical Analysis 2: Comparison: Behavioral & Environmental Intervention (BEI) vs Attention Placebo Group (API); Test type: Superiority or Other; p = .77, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Adherence to Beta Blockers
Description: as for outcome 1
Time Frame: 6 months from baseline
Measure: Median (Inter-Quartile Range); unit: proportion of refill compliance
Arm/Group | Comprehensive Behavioral Intervention (BI) | Behavioral & Environmental Intervention (BEI) | Attention Placebo Group (API)
Number analyzed (Participants) | 28 | 22 | 24
proportion of refill compliance | 0.95 [0.83 to 1.0] | 0.97 [0.76 to 1.0] | 1.0 [0.99 to 1.0]
Statistical Analysis 1: Comparison: Comprehensive Behavioral Intervention (BI) vs Attention Placebo Group (API); Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney) — For this pilot study, the type 1 error was set at 5%
Statistical Analysis 2: Comparison: Behavioral & Environmental Intervention (BEI) vs Attention Placebo Group (API); Test type: Superiority or Other; p = .06, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Self-reported Medication Adherence
Description: Assessed using Morisky medication-taking scale. Higher score corresponds to worse adherence.
Time Frame: 6 months from baseline
Measure: Number; unit: participants
Arm/Group | Comprehensive Behavioral Intervention (BI) | Behavioral & Environmental Intervention (BEI) | Attention Placebo Group (API)
Number analyzed (Participants) | 27 | 29 | 30
participants
  Low adherence | 2 | 4 | 1
  Medium adherence | 9 | 11 | 8
  High adherence | 16 | 14 | 21
Statistical Analysis 1: Comparison: Comprehensive Behavioral Intervention (BI) vs Attention Placebo Group (API); Test type: Superiority or Other; p = 0.60, Fisher Exact — For this pilot study, type 1 error was set at 5%
Statistical Analysis 2: Comparison: Behavioral & Environmental Intervention (BEI) vs Attention Placebo Group (API); Test type: Superiority or Other; p = 0.16, Fisher Exact

ADVERSE EVENTS:
Groups:
- Arm 1: Comprehensive behavioral intervention (BI) - Participants will receive the BI that is based on the transtheoretical model, which targets stage of change, decisional balance and self-efficacy, while also assessing and counseling regarding the barriers and facilitators of HF care, and to improve self-regulatory care such as self-monitoring, self-evaluation, feedback and reinforcement.
  Telephone-Delivered BI: Behavioral Intervention will be delivered over the phone.
- Arm 2: Behavioral & Environmental Intervention (BEI) - Participants in this arm will receive the BI but will also receive environmental tailoring. Environmental Tailoring consists of Built Environment Tailoring (BET) where the intervention will incorporate aspects from the patients' environment, such as accessibility of health food stores or recreational facilities. Environmental Tailoring also consists of Human Environment Tailoring (HET) which incorporates patients' social support. Caregivers will be enrolled for patients in this arm of the study and they will also receive health education.
  Telephone-Delivered BEI: Behavioral and Environmental Intervention will be delivered over the phone
- Arm 3: Attention Placebo Group (API) - patients will receive non-tailored counseling on general health topics.
  Telephone-Delivered API: Attention Placebo Intervention will be delivered over the phone
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 6/33 | 1/33 | 3/33
Other Adverse Events (participants affected / at risk) | 4/33 | 0/33 | 3/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=33) | Arm 2 (N=33) | Arm 3 (N=33)
Death (General disorders) | 2 (2) | 0 (0) | 2 (2)
Cancer (General disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Hospital admission for heart failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=33) | Arm 2 (N=33) | Arm 3 (N=33)
coronary artery bypass graft (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
angina (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Broken bones (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Torn ligament (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes